CLINICAL TRIAL: NCT06486766
Title: InfluSMS: Effectiveness of SMS Nudging to Increase Coverage of Influenza Vaccination Among Elderly From the Majority Population, and Among Elderly From Immigrant Groups With Low Vaccination Coverage
Brief Title: Effectiveness of SMS Nudging to Increase Coverage of Influenza Vaccination Among the Elderly
Acronym: InfluSMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Oslo (Other); Finnish Institute for Health and Welfare (Other Government); University of Turku (Other); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 30052
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-06

CONDITIONS: Influenza
Keywords: influenza vaccination; adult vaccination; coverage; uptake; behavioral nudging; vaccine hesitancy; undervaccination; migrant health
MeSH Terms: conditions — Influenza, Human; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: The trial is conducted in three populations of elderly (aged 65 years or older) residing in Norway: (i) the general population; (ii) immigrants born in Poland; (iii) immigrants born in Ukraine. In all three populations, the control arm is standard care, i.e., no individual reminder for influenza vaccination. All populations have an intervention arm that will receive an SMS nudge in the Norwegian language. In addition, the Polish and Ukrainian immigrant populations include a second intervention arm that will receive an SMS nudge in Polish or Ukrainian, respectively.
Who Masked: Outcomes Assessor
Masking Description: The outcome measure of the trial is based solely on routinely collected data and those reporting/registering this information will not be aware of whether a vaccinated individual has received an SMS nudge. Thus, the trial is blinded to the outcomes assessor. Moreover, treatment allocation is randomized and computer-generated, there is no interaction between the InfluSMS project team and study participants, and the InfluSMS researchers work with de-identified data and do not know the identity of any participant in the dataset. Due to the inherent characteristics of the intervention, treatment allocation cannot be blinded for participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standard care: Influenza vaccination is generally recommended to all individuals aged 65 or older, but there is no systematic individual invitation/reminding/scheduling for vaccination by SMS or any other mode. The control arm is applicable to all three populations (general population, immigrants born in Poland, immigrants born in Ukraine)
- Norwegian SMS (Experimental)
  Interventions: Behavioral: Norwegian SMS
- Polish/Ukrainian SMS (Experimental)
  Interventions: Behavioral: Polish/Ukrainian SMS

INTERVENTIONS:
Behavioral: Norwegian SMS — Individuals receive a SMS in Norwegian language at the start of the influenza season, to remind them they are recommended to get the influenza vaccine. This intervention arm is applicable to all three populations (general population, immigrants born in Poland, immigrants born in Ukraine)
  Arms: Norwegian SMS
Behavioral: Polish/Ukrainian SMS — Individuals receive an SMS in the official language of their native country (i.e., Polish or Ukrainian) at the start of the influenza season, to remind them they are recommended to get the influenza vaccine. This intervention arm is only applicable to the two immigrant populations (immigrants born in Poland, immigrants born in Ukraine)
  Arms: Polish/Ukrainian SMS

SUMMARY:
The trial will investigate to what extent SMS reminders for influenza vaccination increases coverage of influenza vaccination among elderly from the majority population, and among elderly from immigrant groups with low vaccination coverage

DETAILED DESCRIPTION:
Background: The coverage of influenza vaccination among elderly in Norway is insufficient, especially in some immigrant groups. To improve public health, there is a need for an intervention that can increase influenza vaccination coverage. Further, interventions tailored to reduce potential barriers among immigrants can reduce health inequities.

Objective: InfluSMS aims to determine if SMS nudging increases vaccination coverage among those aged 65 or older (i) in Norway's general population; (ii) among immigrants born in Poland; (iii) among immigrants born in Ukraine; and to evaluate the impact of SMS nudging in Norwegian versus in the official language of the native country of immigrants born in Poland or Ukraine.

Methods: InfluSMS is a pragmatic randomized controlled trial conducted among people aged 65 or older residing in Norway. Influenza vaccination coverage is the main outcome, measured in control and intervention arms for each of the three populations listed above. In all three populations, the control arm is standard care, i.e., no individual reminder for influenza vaccination. All populations have an intervention arm that will receive an SMS nudge in the Norwegian language. In addition, the Polish and Ukrainian immigrant populations include a second intervention arm that will receive an SMS nudge in Polish or Ukrainian, respectively. Allocation to study arm is randomized, and the intervention will take place at the start of the 2025/2026 influenza season. All eligible individuals will be passively followed up through the National Immunisation Registry SYSVAK, from which individual influenza vaccination status three months after the SMS nudge will be extracted.

Results: Inclusion of participants will start in the third quarter of 2025, and the registry data will be available in the first quarter of 2026. Coverage rates of each strategy, and coverage differences between strategies will be presented.

Implications: SMS nudging could be integrated into the national influenza vaccination program if the trial shows it effectively increases influenza vaccination coverage among the elderly. Further, the trial will establish whether language is a barrier for influenza vaccination uptake among recent immigrant groups that have low influenza vaccination coverage, and to what extent this potential barrier can be diminished by SMS nudging in the official language of their native country.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65+ (age at the end of 2025, i.e., born 1960 or earlier)
* Resident in Norway and have a valid ID number on 1 September 2025
* Have a registered mobile phone number

Exclusion Criteria:

* Have received the 2025 influenza vaccine prior to the SMS nudge dispatch date
* Have emigrated or died before SMS nudge dispatch date

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination coverage (%) | Three months following the intervention, during the 2025/2026 influenza season
  The percent uptake of the influenza vaccine in the population of interest

OTHER OUTCOMES:
COVID-19 vaccination coverage (%) | Three months following the intervention, during the 2025/2026 influenza season
  The percent uptake of the COVID-19 vaccine in the population of interest

CONTACTS AND LOCATIONS:
Overall Officials: Bo T Hansen, PhD, Principal Investigator — Norwegian Institute of Public Health

IPD SHARING:
Plan to Share IPD: No
The project is not allowed to share the data. Data access requires legal permissions and applications for data must be directed to the registries involved

REFERENCES:
- [Derived] Hansen BT, Klungsoyr O, Labberton AS, Saaksvuori L, Rydland KM, Odeskaug LE, Wisloff T, Meijerink H. Effectiveness of Text Messaging Nudging to Increase Coverage of Influenza Vaccination Among Older Adults in Norway (InfluSMS Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 25;14:e63938. doi: 10.2196/63938. PMID 39998878